CLINICAL TRIAL: NCT05190341
Title: Ibuprofen Versus Ketorolac for Pain Relief During Hysterosalpingogram
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB voted to terminate the protocol for noncompliance
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 221063
Record Dates: First submitted 2021-10-29; First posted 2022-01-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Infertility, Female
Keywords: hysterosalpingogram; ibuprofen; ketorolac
MeSH Terms: conditions — Infertility, Female | interventions — Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial- 88 sequential patients randomized to receive either ibuprofen on ketorolac 1 hr before HSG
Who Masked: Participant, Care Provider, Investigator
Masking Description: Research pharmacist has provided either 800mg ibuprofen or 30mg ketorolac into oral capsules, and randomized sets of pills in packages 1-88. Research physicians and patients blinded which pill sets contain which drug. Will be revealed after data collection complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Experimental): Patients randomized to this arm will receive an identical capsule to the other patient arm, and receive 800mg ibuprofen 1 hour before HSG.
  Interventions: Drug: Ibuprofen 800 mg oral
- Ketorolac (Experimental): Patients randomized to this arm will receive an identical capsule to the other patient arm, and receive 30mg ketorolac 1 hour before HSG.
  Interventions: Drug: Ketorolac 30mg oral

INTERVENTIONS:
Drug: Ibuprofen 800 mg oral — 1 hour before HSG
  Other Names: Advil; Motrin
  Arms: Ibuprofen
Drug: Ketorolac 30mg oral — 1 hour before HSG
  Other Names: Toradol
  Arms: Ketorolac

SUMMARY:
Hysterosalpingogram (HSG) testing is a vital part of the workup for infertility patients. It is often noted to be biggest pain that patients undergo during the workup. Several studies have attempted to find a therapy that reduces pain, with non-steroidal anti-inflammatory drugs such as oral ibuprofen the current mainstay. Our study attempts to determine which of the following NSAIDS is best at reducing pain associated with the HSG procedure: oral ibuprofen versus oral ketorolac .

DETAILED DESCRIPTION:
Describe step-by-step how the study will be conducted from beginning to end

1. After IRB approval, the research pharmacist will provide motrin and ketorolac in identical packets labeled 1-88, after receiving the randomization strategy/number set from the research monitor.
2. REI physician on the protocol will screen patient for inclusion/exclusion from study at new patient consult or at future follow up visit when need for HSG is decided.
3. If patient pt screens eligible, discuss study. If elects participation then consent patient and randomize to group.
4. At time of scheduling HSG, patient will need to remind nursing that they are in HSG study. Nursing should also have the list of patients to reference when scheduling HSGs. Patients in the study will need to check in at the REI clinic 70 minutes prior to HSG in order to take their meds 60 minutes prior to scheduled procedure time. At same visit, REI RN will perform urine pregnancy test as previously scheduled.

   a. meds will be kept in a locked cabinet in the REI research office in opaque sealed envelopes.
5. Patient will then go check into Radiology for their HSG.
6. HSG will be performed per standard clinical protocol. The HSG will be performed by REI physicians and OB/GYN residents (who are rotating on REI), which are the current standard of practice.
7. A nurse or provider associated with the study will need to be at the HSG for the sole purpose of study assistance. The provider performing the HSG, the study personnel recording pain levels, and the fluro tech will not be aware of the type of pre-procedural medication the patient received. The nurse or provider of study personnel will do the following:

   1. time the procedure from placement of speculum through deflation of catheter balloon and removal of catheter. Record time in seconds (can write mins:seconds and then convert later).
   2. record who performed the procedure, if a tenaculum had to be used, and if an attending had to take over the procedure
   3. help patient record pain scale marks on the VAS sheet at the designated time periods.

7. For clarity- there will be at least three providers at each HSG for study enrolled patients.

1. A provider who does the HSG
2. A fluoro technician to capture fluoro images for teh HSG
3. A study affialitied person to record pain scores for patient as above 8. At the conclusion of study recruitment, the blinded researchers will gain access to the subject ID's cohort status (ibuprofen vs ketorolac), and study analysis will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* premenopausal females age 18-45
* patients currently undergoing HSG as part of routine work-up for infertility or subfertility, - - patients with negative urine pregnancy test within 24 hours of the scheduled procedure
* patients having performance of HCG between menstrual cycle days 5-12n

Exclusion Criteria:

* Non-English speaking
* patients with history of previous HSG performed
* patients with contrast allergy or other contraindications to HSG
* patients with contraindications to NSAID use
* Patients with the following:
* unwilling to consent
* positive urine pregnancy test within 24 hours of the scheduled procedure
* active renal or hepatic disease
* chronic narcotic users
* use of pain medications within 12 hours of the scheduled procedure
* patients with chronic pain conditions (fibromyalgia, complex regional pain syndrome, etc.)
* patients with unknown uterine anatomical pathology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Pain during contrast infiltration | Between 0 seconds and 5 minutes
  Pain on Visual Analogue Scale (0-100)

SECONDARY OUTCOMES:
Pain at baseline (before procedure start) | Between 0 seconds and 5 minutes
  Pain on Visual Analogue Scale (0-100)
Pain with HSG catheter placement | Between 0 seconds and 5 minutes
  Pain on Visual Analogue Scale (0-100)
Pain at completion of HSG | Between 0 seconds and 5 minutes
  Pain on Visual Analogue Scale (0-100)
Pain 5 minutes following HSG | 5 minutes after procedure
  Pain on Visual Analogue Scale (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Pier, Principal Investigator — Madigan Chief of REI, Department of OBGYN
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No